CLINICAL TRIAL: NCT06345859
Title: Ambulatory Phenotyping With Real-Time Indices of Discordant Affect Regulation: Exploring Opportunities for Targeted Intervention in Depression
Brief Title: Regulation of Affect and Physiology in Depression
Acronym: RAPID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jonathan Stange, Assistant Professor of Psychology and Psychiatry & the Behavioral Sciences, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UP-23-00467; R01MH133842 (NIH)
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osc+ (Experimental): Osc+ condition. In the Osc+ condition, participants will see an on-going record of their heart rate over time. They will be instructed to engage in paced breathing and to try to maximize their oscillation score. The paced breathing will be adapted to a rate that allows them to maximize their high amplitude heart rate oscillations.
  Interventions: Behavioral: Heart rate variability biofeedback
- Osc- (Active Comparator): Osc- condition. In the Osc- condition, participants will also see an on-going record of their heart rate over time, and will be instructed to engage in paced breathing. However, they will be asked to try to keep their heart rate steady and avoid oscillations and will get points on an 'alertness' score that inverts the Osc+ 'oscillation' score.
  Interventions: Behavioral: Heart rate variability biofeedback

INTERVENTIONS:
Behavioral: Heart rate variability biofeedback — This is a Phase 2 parallel intervention design with random assignment. We will randomly assign participants to one of two biofeedback conditions. Both conditions involve completing breathing exercises at home, 30 minutes per day for 10 days, while receiving continuous feedback about parasympathetic activity from the computer.

SUMMARY:
Although treatments for depression are effective for many people, not everyone responds to treatment. This lack of treatment response could be due, in part, to the presence of multiple underlying causes of people's depression. This study aims to identify subtypes of depression, based on two factors: how successful people perceive themselves to be at regulating their affect in everyday life; and how much activity in the parasympathetic nervous system increases during moments when people try to regulate. The study involves ambulatory assessment of affect, regulation strategies, and physiological activity in everyday life, in a sample of young adults with remitted major depressive disorder and healthy volunteers. We will study regulation responses in the lab to further determine how subtypes differ in neural, physiological, and behavioral responses. Finally, participants will be randomly assigned to a remote, self-administered biofeedback intervention (vs. control intervention) designed to increase parasympathetic activity and physiological regulation success. While engaging in biofeedback at home for 10 days, participants will simultaneously repeat the ambulatory assessments. This design will allow us to determine the proximal impact of biofeedback on indices of regulation success in everyday life, and whether biofeedback has differential impact on regulation success for different subtypes.

ELIGIBILITY:
Inclusion Criteria for Participants with Remitted Depression:

1. Age 18-27.
2. Meeting criteria for lifetime major depressive disorder.
3. Currently meeting criteria for full remission (absence of clinically significant symptoms) for at least eight weeks, and having a Hamilton Depression Rating Scale score of less than or equal to 7.

Inclusion Criteria for Healthy Volunteer Participants:

1. Age 18-27.
2. No lifetime history of any psychiatric disorder.
3. No first-degree relatives with a mood disorder.

Exclusion Criteria (same for all participants):

1. Change in psychotropic medication use within the last 30 days
2. Autism spectrum disorder
3. Current eating disorder
4. Intellectual disability
5. Substance use disorder within the past 6 months
6. Contraindications for magnetic resonance imaging or electrocardiogram assessment (e.g., presence of metal in body, claustrophobia, cardiac device, pregnancy).

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 252 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Physiological regulation success | The two 10-day ambulatory assessment periods.
  A slope representing the strength of the relationship between how much each individual's heart rate variability increases after engaging in adaptive regulation strategies (reappraisal, distraction, and/or acceptance). Values of this variable during the 10-day biofeedback intervention period will be compared to values during the 10-day baseline ambulatory assessment periods.
Average level of heart rate variability | The two 10-day ambulatory assessment periods.
  An intercept representing the average level of heart rate variability each person experienced. Values of this variable during the 10-day biofeedback intervention period will be compared to values during the 10-day baseline ambulatory assessment periods.

SECONDARY OUTCOMES:
Perceived regulation success | The two 10-day ambulatory assessment periods.
  An intercept representing the average degree of success each person perceived in regulating their affect. Values of this variable during the 10-day biofeedback intervention period will be compared to values during the 10-day baseline ambulatory assessment periods.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Per our data sharing plan, we plan to share the de-identified final research data with the broader scientific community via the National Institute of Mental Health Data Archive. This includes fMRI data, ambulatory data, and clinical, behavioral, and self-report measures.